CLINICAL TRIAL: NCT01562353
Title: A Pilot Study to Determine the Genetic Biomarkers Predictive of the Development of Prescription Opioid Addiction in Patients Treated for Pain Using a Comparative Transcriptomic Analysis of Gene Expression in Peripheral Blood Cells
Brief Title: Determining Genetic Biomarkers Predictive of the Development of Prescription Opioid Addiction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Analgesic Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: CPH.CSA.0005
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Usage of Prescription Opioids
Keywords: Opioid Dependence; Opioids for the treatment of pain
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — One tube (2.5-5.0 mL) of blood will be drawn from each subject during the visit for mRNA testing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Subject has a diagnosis of current prescription opioid dependence (confirmed by the MINI). Subject had no history of dependence on alcohol or illicit or prescription drugs, including opioids, prior to prescription opioid exposure for the treatment of chronic pain.
- Control: Subject's prescribing physician has reported absence of significant problematic behavior with respect to prescription opioids or other substances while under the physician's care. Subject has a negative urine drug screen for alcohol, illicit drugs, and nonprescribed controlled substances at screening. Subject has no current or past substance abuse or dependence (confirmed by the MINI and medical history).

SUMMARY:
This is a clinical study on patients who have been prescribed opioids (narcotic pain relievers) for the treatment of pain, to determine what genetic factors influence outcome of treatment. Procedures include: an initial telephone prescreening, completion of a number of questionnaires, and a blood draw to determine genetic factors. Participants will take part in a one-time clinic visit, during which all procedures will be completed.

The investigators hypothesize that several classes of genes, including genes in opioid, pain, and reward pathways, will differentiate opioid-dependent subjects from opioid-exposed nondependent subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older.
* Subject is willing and able to speak, read, and write in English and comply with all study procedures.
* Subject is willing and able to voluntarily sign and date an Informed Consent Form (ICF), approved by an Institutional Review Board (IRB), prior to the conduct of any study-specific procedures.
* Subject has been prescribed opioids for the treatment of pain for at least 6 months at the time of the study.

Cases:

* Subject has a diagnosis of current prescription opioid dependence (confirmed by the MINI).
* Subject had no history of dependence on alcohol or illicit or prescription drugs, including opioids, prior to prescription opioid exposure for the treatment of chronic pain. Patients who have abused these substances but have not met criteria for dependence (confirmed by the MINI and/or medical history) will be included.

Controls:

* Subject's prescribing physician has reported absence of significant problematic behavior with respect to prescription opioids or other substances while under the physician's care.
* Subject has a negative urine drug screen for alcohol, illicit drugs, and nonprescribed controlled substances at screening.
* Subject has no current or past substance abuse or dependence (confirmed by the MINI and medical history).

Exclusion Criteria:

* Subject has any condition that poses undo study-related risk, or that interferes with assessment.
* Subject is not willing to have blood drawn or has any condition that in the investigators' opinion precludes having blood drawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of 15 subjects per group will be sought. Cases and Controls will be selected by a community-based advertising program supplemented by referrals from clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
mRNA Levels | 1 day
  mRNA levels for all known genes and exons

SECONDARY OUTCOMES:
FTQ | 1 day
  Family Tree Questionnaire
TEQ | 1 day
  Trauma Exposure Questionnare
LSQ | 1 day
  Life Stress Questionnaire
POCS | 1 day
  Prescription Opioid Craving Scale
POAQ | 1 day
  Prescription Opioid Analgesic Questionnaire
mARCI | 1 day
  Modified Addiction Research Center Inventory
MINI | 1 day
  Mini International Neuropsychiatric Interview

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel P Katz, MD, MS, Principal Investigator — Analgesic Solutions
Locations (1):
- Analgesic Solutions, Natick, Massachusetts, United States